CLINICAL TRIAL: NCT04928963
Title: Phase I/II Randomized Clinical Study of Cycles of a New Formulated FMD in Prefrail Elderly.
Brief Title: Fighting Immunosenescence and Promoting Immunity by a Fasting-mimicking Diet Elderly.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Alessio Nencioni, Full Professor, University of Genova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FAIS
Record Dates: First submitted 2021-06-11; First posted 2021-06-16 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Frailty; Inflammation; Immune System Disorder
Keywords: nutritional status; fasting; fasting-mimicking diet; immunosenescence
MeSH Terms: conditions — Frailty; Inflammation; Immune System Diseases; Fasting

STUDY DESIGN:
Intervention Model Description: This is a pilot, double arm prospective trial assessing feasibility and safety of a 5-day fasting-mimicking diet in pre-frail elderly patients who are going to be vaccinated against flu. Patients will be randomized for FMD or for placebo diet and both of the groups will recieve flu vaccine.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fasting mimicking diet (Experimental): Fasting mimicking diet will be provided with all food to be consumed during each of the 2 cycles. The components of the diet will be approximately 30% calorie restricted and 50% protein restricted but supplemented with 50% of the RDA in vitamins and minerals and also supplemented with both nonessential and essential amino acids identified in animal studies to be effective.
  Interventions: Dietary Supplement: Prolon - FMD
- Placebo diet (Placebo Comparator): One meal which substitute or lunch or dinner for 5 days, without calories restriction.
  Interventions: Dietary Supplement: Prolon - FMD

INTERVENTIONS:
Dietary Supplement: Prolon - FMD — Prolon by L-Nutra is a medically-designed dietary kit providing the food to eat for five days. Day 1 of Prolon provides ~4600 kJ (11% protein, 46% fat, and 43% carbohydrate), whereas days 2-to-5 provide ~3000 kJ (9% protein, 44% fat, and 47% carbohydrate) per day.

SUMMARY:
Background: Immunosenescence is an aging-dependent phenomenon underlying age dependent deterioration in the function of the immune system, characterized by a decline in B and T cells with a relative increase in natural killer (NK) cells. Aging also promotes chronic inflammation accompanied by increased levels of pro-inflammatory cytokines. Both immunosenescence and inflammation contribute to frailty, which is a geriatric syndrome characterized by age-related deterioration in multiple physiological systems resulting in greater vulnerability to stressors and increased risk of poor outcomes including longer hospital stays, postoperative complications, poor responses to vaccination, functional decline, and death.

Although pharmacological interventions could be developed to address immunosenescence, inflammation and frailty, a dietary intervention that does not cause weight or muscle loss may be a preferable option, particularly if it is periodic in nature and it only needs to be adopted for a few weeks per year.

Hypothesis: We will test the hypothesis that a newly formulated and relatively high calorie fasting mimicking diet (FMD) to be administered to subjects age 65-80 once a month for 5 days for two to six cycles can partially reverse immunosenescence and inflammation, thus contributing to the reduction of frailty.

Aims: This proposal is divided into 2 main tasks:

Task 1: We will determine whether FMD cycles in mice: a) prevent frailty syndrome onset and symptoms B) delay or reverse age-related immunosenescence and inflammaging, C) improve the functionality of bone marrow cells, D) enhances the response to flu vaccination. Task 2: A )We will develop a special relatively high calorie FMD medical food for testing in humans, B) We will test the safety and efficacy of the FMD medical food in an aged and frail individuals (65-80 yr) for 2-5 day cycles preceding their annual influenza vaccination. Expected results: In mice, we expect that the FMD diet will reduce the clinical signs of frailty during aging, and in particular increase immune system influenza vaccine response by preventing immunesenescence. We expect that the FMD will reduce phosphorylation of mTOR and of its downstream targets, and induce autophagy and apoptosis in WBCs. These effects are anticipated to remove damaged cells and promote the activation of hematopoietic stem cells and the generation of new WBCs. We also expect that the transient increase in corticosteroids and removal of damage immune cells will be accompanied by a decrease in systemic inflammation. Increased performance on rotarod and other measures of frailty is also anticipated. In humans, we expect that the FMD will be well tolerated by the pre-frail elderly without major adverse events and that it will be possible to achieve high compliance to this diet. We also anticipate that elderly undergoing the FMD protocol followed by 30 days of a normal diet plus supplements will exhibit better functional status and better response to the flu vaccine as compared to patients from the control arm. An improvement in handgrip strength and in lean body mass, as detected by BIA, is also expected, at least in a fraction of the patients from the intervention arm. Impact: Frailty is a geriatric syndrome characterized by age-related deterioration in multiple physiological systems and homeostatic mechanisms, resulting in greater vulnerability to stressors and increased risk of poor outcomes including longer hospital stays, postoperative complications, poor responses to vaccination, functional decline, and death. Thus, the identification of a dietary strategy, potentially to be applied for only 10 days a year but able to rejuvenate the immune profile and function while reducing systemic inflammation could have a major impact on both healthspan and health-related expenses. Because older individuals are often taking multiple drugs, the dietary intervention being investigated here would also reduce the potential toxicity of an additional pharmacological intervention.

DETAILED DESCRIPTION:
A phase I/II randomized clinical study will be performed to assess feasibility, safety, and efficacy (improvement of the response to vaccination, but also functional status improvement or maintenance) of two cycles of FMD (1 week) administered 30 days apart, preceding flu vaccination in pre-frail elderly subjects. The study will enrol 40 pre-frail subjects aged 65-80 years. Subjects will be excluded if they have known immunosuppressive disorders or medications or have not received influenza vaccination in the previous two years. Subjects will be randomized 1:1 to Arm A (FMD) or Arm B (regular diet). Subjects in Arm A will receive the 5 day FMD diet once a month for 2 months (2 cycles completed in 40 days: 5-30-5).

This is based on the regimen adopted in our ongoing study with younger subjects but involves one less cycle to minimize weight loss, and other potential side effects in elderly subjects. The primary endpoint will be diet safety: the side effects of the diet will be assessed by weight change, headaches, blood pressure, and by closely monitoring body composition, i.e. lean body mass, by bio-impedance measurements, handgrip strength and DEXA scans. The secondary endpoints will include: i) the compliance with the FMD; ii) the improvement of frailty parameters and prevention of disability in patients 65-80 years of age; iii) the improvement in immune parameters after 2 cycles of the diet and will be based on measures of improved T cell response, reduced inflammation, improved lymphoid/myeloid ratios and HSC/pre-HSC number, improved B cell numbers and CSR; iv) the efficacy of the influenza vaccine assayed by higher antibody titer levels. In addition, we will also document the number of flu episodes over the course of the trial. The trial will be carried out over a period of 3 years and all subjects will be vaccinated in the fall of each year with the current preparation of the inactivated virus influenza vaccine (Fluzone® high dose, Sanofi Pasteur Inc.) at the San Martino Hospital. During the flu season each participant will receive weekly reminders to call in and report any influenza like symptoms. These will include respiratory symptoms (cough, sore throat, shortness of breath and nasal stuffiness) and systemic symptoms (headache, malaise, fatigue, fever or feverishness and muscle aches). Flu-like illnesses will be documented based on the report of two respiratory symptoms or one respiratory and one systemic symptom when influenza is known to be circulating in the local community. A laboratory diagnosis of influenza illness will be confirmed from the results of nasopharyngeal swabs for virus culture, and/or a pre- to post-illness 4-fold or greater rise in antibody titer. Blood samples will be collected at baseline, after 2 diet cycles prior to vaccination and at 4 weeks after vaccination. The study period for this trial will be 2-5 day diet cycles (5-30-5) followed by a single flu vaccination per year. Each diet cycle will consist of 5 days of FMD followed by 30 days of the subjects' usual diet plus a plant-based daily protein and fat supplement (20 grams of proteins + 30 grams of olive oil and 30 grams (total) of walnuts, hazelnuts and almonds). This daily supplement serves at minimizing weight loss caused by the 5 day FMD. At the first visit, subjects will undergo a physical evaluation to assess health and frailty status, and medical history will be noted. Blood samples will be collected for baseline measurements.

Subjects in the FMD arm will be given a 2 cycle supply of the diet with instructions. Before receiving the second FMD cycle, patients will undergo a second physical examination at the geriatrics Clinic of the University of Genoa which will include the assessment of body composition and the administration of the second FMD cycle will only be allowed in the absence of a decrease in lean body mass (vs. baseline) as detected by BIA, handgrip strenght and by DEXA. Two weeks after completion of second diet cycle, subjects will return for physical evaluation, blood collection and vaccination. The third and final visit will be 4 weeks following vaccination, the subjects will undergo a physical evaluation and assessment of body composition and blood samples will be collected. At this visit, subjects will also be instructed to call the research coordinator to report malaise, discomfort, influenza or respiratory symptoms. Further follow-up will be over the phone to monitor onset of influenza. Nasopharyngeal swabs for virus culture and confirmation of influenza will be collected if possible within 72 hours of a subject reporting symptoms of influenza. DIET: Subjects randomized to the restricted diet arm (A) will be provided with all food to be consumed during each of the three cycles. The exact components of the diet will depend on results obtained in Task

1 but the diet is anticipated to be approximately 30% calorie restricted and 50% protein restricted but supplemented with 50% of the RDA in vitamins and minerals and also supplemented with both nonessential and essential amino acids identified in animal studies to be effective. Amino acid supplementation levels will depend on published clinical studies demonstrating safety and will not exceed the recommended daily levels. Subjects in the control arm will receive dietary advice per the standard practice of the treating physician. This will include consultation with a registered dietitian. A major focus will be placed on ensuring that subjects do not lose weight (unless obese at baseline) nor lose lean body mass. They will also be asked to maintain a diary of the food consumed and approximate amounts.

VACCINATION: Subjects will be vaccinated with the standard dose of the Fluzone® high dose vaccine from Sanofi Pasteur Inc. for each year. This vaccine has four times the normal antigen contained in the regular flu vaccine and is specially designed for individuals 60 and older.

Criteria for Removal from Study:

Subjects will be removed from the study if they do not receive the vaccination Subjects will be removed from study if they have unacceptable toxicity related to the diet.

Subjects will be removed from study is they are unable to regain at least 95% of their body weight after the first and 92% after the second cycle. Subjects will be removed from study in the presence of a decrease in bioimpedance phase angle exceeding 5% of the baseline value or whenever the phase angle will drop below 5°; or, alternatively, in those patients in which bioimpedance measurements were unreliable/unattainable, in the presence of a decrease in handgrip strength or in lean body mass detected by DEXA >5% of the baseline value. Subjects may voluntarily withdraw from the study at any time, for any reason. STUDY OBSERVATIONS Visit 1: A complete medical history will be documented at the first visit at the San Martino Hospital (Prof.

P. Odetti, MD, Prof. A. Nencioni). This will include documentation of chronic diseases and any diseases that could increase risk for influenza including congestive heart failure, ischemic heart disease, chronic lung disease, diabetes, kidney failure, neoplastic disorders and immune dysfunction weight and performance status. All medications will be recorded. A physical will be performed, and Body Mass Index (BMI) and body composition will be determined and must be within inclusion parameters. Pre-frailty will be diagnosed in participant whether one or two of Fried modified criteria for frailty will be present. A blood draw will be performed. Baseline laboratory measurements will include a CBC, glucose, ketone bodies, insulin, IGF-I, IGFBP-1, cytokine panel, lymphoid/myeloid ratio, CD4+/CD8+ ratio, naïve/ memory T cells ratio and CD8+CD28+ T cells. To assess humoral immunity, percentages and absolute numbers of CD19+ B cells, naïve, IgM memory and switch memory B cells will be assessed. Briefly, PBMC's isolated from whole blood will be enriched for CD19+ B cells using anti-CD19 Microbeads (Miltenyi Biotech). To isolate naïve, memory and switch memory cells, CD19 cells will be sorted using a flow cytometer after staining with PE-conjugated anti-CD27, biotin-SP-conjugated ChromPure human IgG, and 20 μl biotin-SPconjugated ChromPure human IgA. To detect CSR in vitro, CD19 B cells will be cultured with anti CD40 and IL-4 for 6-7 days. AID expression in the stimulated B cells will be measured by RT-PCR. E47 expression will be measured by western blot. Visit 2: Subjects will return to the clinic upon completion of one cycle of the diet. The participants will be subjected to a new medical examination to evaluate their physical activity, neuropsychological and to determine the frailty index. In addition, they will also undergo a body composition assessment by bioimpedance measurement, by DEXA scan and by handgrip strength. A blood draw will be performed.

Laboratory values will include all measurements as above to assess post-diet changes in all the parameters described above. Visit 3 (two weeks after the second FMD cycle): same as in visit 2. In addition, all subjects will receive a single injection of influenza vaccination. Visit 4: Subjects will return at 4 weeks post vaccination, when antibody titers are expected to peak. We will perform the clinical examinations and the body composition assessments performed on previous visits on the participants. Laboratory measurements will be as above. In addition, antibody titers in serum will be measured by the haemagglutination inhibition assay. Hemagglutinin for each virus strain will be obtained from the CDC stock. 2 fold dilutions of serum from 1/10 to 1/1024 will be used. Chronic agerelated muscle loss affects >30% of individuals over 60 and >50% of individuals over 80. Insufficient protein intake in the elderly may promote loss in muscle mass by preventing muscle protein synthesis. Thus, bioimpedance measurements and whole body DEXA scans will be conducted in order to ensure that the diet does not cause loss in muscle mass. Follow-up: The subjects enrolled in the study will be called every three months after the fourth visit (see above) to undergo physical and psychological examinations in order to evaluate the FMD efficacy in preventing frailty, reinforcing the immune system and increasing efficacy of influenza vaccine. During the predicted influenza season in the local area, subjects will receive weekly phone calls from the trial coordinator to document any symptoms and to remind them to call in to report symptoms. If possible NP swabs will be collected within 72 hours of reporting of symptoms by having the RN travel to the subjects homes. The incentive for participants to report symptoms early will be access to free diagnosis and referral to the primary physician for treatment of influenza illness. Non-compliance will be defined as consumption of <50% of the prescribed diet and/or consumption of >150 kcal non-prescribed food on any of the days of the FMD. Results for subjects with less than a 50% reduction in IGF-I and 40% reduction in glucose compared to baseline will be analyzed (intention-to-treat) but a secondary analysis excluding these patients (suspected of being non-compliant) may be performed.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants are age 65-80 who may have underlying chronic diseases but no advanced kidney disease or diabetes requiring insulin.
2. Subjects with a diagnosis of pre-frailty according to Fried's modified criteria.
3. Subjects with a minimum BMI of 20 kg/m2
4. Subjects with a bio-impedance phase angle >5°.

Exclusion Criteria:

1. Known allergy to components of the kit.
2. A previous significant reaction to vaccination or if they refuse to receive influenza vaccination.
3. Known immunosuppressive disorders or medications;
4. Subjects who report respiratory illness within the two-week period prior to vaccination;

7. Subjects with a BMI <20 8. Subjects with a bio-impedance phase angle <5°.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Safety of FMD in terms of percentage of patients experiencing adverse events and/or worsening of nutritional status | 6 months
  To obtain clinical data on safety of the FMD, in pre-frail elderly (65-80) as assessed by percentage of patients (%) experiencing > grade 3 adverse events and/or a significant decrease in their lean body mass (kg) and/or with a reduction of phase angle <5° assessed with bio-impedance measurements.
Feasibility of FMD in terms of percentage of patients able to complete the diet regimen | 6 months
  To evaluate the feasibility of the FMD in pre-frail elderly (65-80) as assessed by the percentage of patients (%) able to achieve the designated diet regimen.

SECONDARY OUTCOMES:
Efficacy of FMD in terms of immune response after Flu vaccine | 1 month
  To evaluate the efficacy of FMD in term of immune response after flu vaccine, antibody titer against Flu (U/ml) will be assessed after 4 weeks from the injection of flu vaccine.
Efficacy of FMD in terms of prevention of frailty | 6 months
  To evaluate the efficacy of FMD in the prevention of frailty patients will be assessed with 40-item Frailty index (Rockwood, 2008). This tool has a score between 0 and 1, with patients considered to be fit with a Frailty index score ≤ 0.08, pre-frail with a score >0.08 and <0.25 and frail with a score ≥ 0.25. Patients considered frail have an high risk of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Alessio Nencioni, Genoa, GE, Italy

IPD SHARING:
Plan to Share IPD: No